CLINICAL TRIAL: NCT01676363
Title: Pilot Study of Diflunisal in HIV-infected Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Julio Montaner, Dr. Julio Montaner, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11-03547; H11-03547 (Other: UBC/Providence Health Care REB)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: HIV Infection
Keywords: diflunisal; anti-inflammatory agents, non-steroidal; antiviral agents
MeSH Terms: conditions — HIV Infections | interventions — Diflunisal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diflunisal (Experimental)
  Interventions: Drug: Diflunisal

INTERVENTIONS:
Drug: Diflunisal — Open-label diflunisal 500 mg twice daily for 4 weeks

SUMMARY:
Diflunisal is an anti-inflammatory drug (like ASA or ibuprofen) that has been used as a painkiller for 20 years. Recent research shows that it may have an anti-HIV effect in the laboratory. Approximately 20 HIV-infected adults who are not receiving antiretroviral therapy will be given diflunisal by mouth twice daily for 4 weeks, at a dose that has been shown to be safe when used to treat pain. Subjects will be monitored closely for safety and will have frequent blood tests during the study to see if the drug has any effect on the level of HIV in their blood.

DETAILED DESCRIPTION:
Following informed consent, potential subjects will undergo a screening visit to determine study eligibility. Within 2 weeks of screening, they will undergo a Day 1 visit for blood testing. At the Day 8 visit on the following Monday, after study visit procedures have been completed, they will commence taking diflunisal 500 mg twice daily by mouth for 4 weeks (Days 8-36, study treatment period), during which they will be seen once a week for blood tests. Following the last dose of diflunisal which will be taken on the morning of Day 36, they will be seen for blood tests after 1 week off the study drug (Days 43, washout phase), and again for a final visit after 2 weeks off study drug, on Day 50.

Subjects will be instructed to take diflunisal 500 mg by mouth in two doses approximately 12 hours apart (+ or - 1 hour), with or without food. A 2-week supply will be dispensed on Days 8 and 22. Study medication bottles (empty or not) will be returned to the clinic on Days 22 and 36. Pill counts will be performed to assess adherence. Adherence will further be evaluated by measuring diflunisal drug levels in plasma samples collected weekly starting at the baseline visit, and assayed at the end of the study.

After the subject has provided informed consent, a screening visit will be performed including a complete medical history and record of concomitant medications to determine study eligibility. Complete physical exam, CBC, platelet count, serum creatinine and estimated GFR, serum potassium, AST, ALT, total bilirubin, CD4 cell count, and pregnancy test for women of child-bearing potential will be performed at the screening visit and repeated at the final study visit. At each study visit, blood will be drawn for HIV RNA, and a serum sample will be collected and stored for measurement of C-reactive protein (CRP), d-dimer, and possibly other inflammatory biomarkers. Plasma (for diflunisal drug level measurement) and peripheral blood mononuclear cells (PBMC's) will be collected and stored weekly from the baseline visit to Day 50. PBMC's will be frozen and shipped in batches to Eric Verdin, MD at the Gladstone Institute of Virology and Immunology (1650 Owens St San Francisco, CA 94158, USA) for analysis of T cell subsets (naïve, memory CD4 and CD8 T cells) and levels of protein acetylation (histone or other) as a surrogate marker of drug activity. Adverse events and concomitant medications will be recorded at the baseline visit and updated weekly.

After completion of the final study visit, subjects will be compensated for their time in the amount of $500. Subjects who need to discontinue the study early, e.g. due to significant clinical or laboratory adverse events related to the study drug, will receive the full stipend at the end of their participation in the study. Subjects who choose to withdraw from the study early or who are withdrawn for study noncompliance will not be eligible to receive the stipend. Subjects who require ongoing reimbursement for travel expenses to enable them to attend study visits will receive advances on their stipend upon providing receipts for parking, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 19 years or over
2. HIV positive by ELISA and Western blot, at least 3 months prior to screening
3. No antiretroviral therapy within 3 months prior to screening
4. Plasma HIV RNA (viral load) > 2,500 copies/mL at screening
5. Current CD4 cell count >350 cells/mm3 at screening
6. Adequate renal function as demonstrated by eGFR >60 mL/min. at screening

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Any HIV-associated symptom or condition (e.g. nephropathy) for which standard antiretroviral therapy is indicated immediately
3. History of peptic ulcer and/or gastrointestinal bleeding
4. Allergy to ASA, other salicylates, or NSAIDs
5. Currently receiving treatment with an ACE inhibitor, ASA, anticoagulants, antacids containing aluminum hydroxide, cyclosporine, diuretics, systemic glucocorticoids, lithium, methotrexate, or other NSAIDs
6. Significant hepatic impairment or active liver disease - screening AST, ALT, or bilirubin >2.5x upper limit of normal (ULN)
7. Hyperkalemia - screening serum potassium >5.5 mmol/L
8. Anemia - screening hemoglobin <85 g/L

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma HIV RNA level | between baseline and end of 4-week treatment, and between end of treatment and end of 2-week washout
  Plasma HIV RNA changes between baseline and end of 4-week treatment, and between end of treatment and end of 2-week washout

SECONDARY OUTCOMES:
Clinical adverse events including serious adverse events | from screening until final study visit on Day 50
Clinically significant changes in laboratory parameters | between screening and Day 50
  changes in complete blood count (CBC), platelets; serum creatinine, estimated glomerular filtration rate (GFR); AST, ALT, total bilirubin; serum potassium; CD4 cell count
Slope of HIV RNA change | during 4-week treatment and 2-week washout phases
Changes in inflammatory biomarkers | during 4-week treatment and 2-week washout phases
  Changes in C-reactive protein (CRP), d-dimer, possibly other biomarkers
Changes in T cell subsets | during 4-week treatment and 2-week washout phases
  Changes in naïve and memory CD4 and CD8 cells
Changes in protein acetylation (histone or other) in peripheral blood mononuclear cells (PBMCs) | during 4-week treatment and 2-week washout phases

CONTACTS AND LOCATIONS:
Overall Officials: Julio Montaner, MD, Principal Investigator — Providence Health Care/ University of British Columbia
Locations (1):
- Immunodeficiency Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada